CLINICAL TRIAL: NCT06849050
Title: The Influence of Acute Continuous Exercise and Adiposity on Appetite Hormones and Neural Correlates of Visual Food Cues
Acronym: ACECRAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Professor David Stensel, Professor of Exercise Metabolism, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18581
Record Dates: First submitted 2025-02-18; First posted 2025-02-27 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-10

CONDITIONS: Overweight; Obesity
Keywords: Appetite; Obesity; Overweight; fMRI; Neural correlates; Exercise; Oxyntomodulin
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Rest in the laboratory from 08:00 to 13:00. For 30-minutes, participants will be asked to wear a face mask, which will measure their oxygen consumption at rest. Ad libitum energy intake assessed at 11:00 (2.5 hours).
- Exercise (Experimental): Rest in the laboratory from 08:00 to 13:00 apart from 60 minutes of treadmill exercise (walking/jogging) performed between 09:00-10:00 (0.5-1.5 hours). Ad libitum energy intake assessed at 11:00 (2.5 hours).
  Interventions: Behavioral: Acute continuous exercise

INTERVENTIONS:
Behavioral: Acute continuous exercise — Exercise, which will involve 60 minutes of brisk walking, or jogging, at 60% of peak oxygen uptake. Participants will be asked to wear a face mask, which will measure their oxygen consumption during the exercise session.
  Arms: Exercise

SUMMARY:
Exercise increases energy expenditure and impacts appetite and energy intake. Some appetite-related hormones such as oxyntomodulin suppress appetite whilst other hormones such as ghrelin stimulate appetite. This study will investigate whether acute continuous walking/jogging influences these hormone concentrations, and whether exercise-induced changes in the hormones correlate with perceptions of appetite, nutritional intake and brain activity in individuals varying in weight status.

DETAILED DESCRIPTION:
Single bouts of exercise transiently suppress appetite and the orexigenic gut hormone acylated ghrelin and increase anorexigenic gut hormone concentrations including peptide YY (PYY) and glucagon-like peptide-1 (GLP-1). These changes occur without stimulating compensatory increases in appetite and energy intake on the day of exercise resulting in a short-term energy deficit. Oxyntomodulin is another gut-derived hormone that suppresses appetite and increases energy expenditure but the influence of acute exercise on oxyntomodulin concentrations in individuals varying in adiposity status has not been investigated. This study will investigate whether acute continuous walking/jogging impacts circulating oxyntomodulin concentrations in individuals who are lean or living with overweight or obesity. The influence of exercise and adiposity on other hormonal, subjective, sensory and neural correlates of appetite will also be explored.

This study is a cross-over design consisting of four visits: a pre-visit, two main trial visits (exercise and control) and a magnetic resonance imaging (MRI) visit. Participants will undertake a preliminary measures visit (pre-visit) to confirm eligibility, complete questionnaires assessing their health, habitual physical activity and eating behaviours, undergo standard anthropometric measurements (height, weight, and hip/waist circumference) and treadmill exercise tests to determine their peak oxygen uptake.

Main trials will be separated by at least seven days for male participants, whereas female participants will complete the two main trials in the follicular phase (the first seven days) of the menstrual cycle. Participants will arrive at the laboratory after fasting overnight for at least 10 hours (plain water is permitted). Participants will then complete assessments of height, weight and either bioelectrical impedance analysis (main trial 1) or air displacement plethysmography (BOD POD®) (main trial 2). A venous cannula will be inserted for the collection of venous blood samples at 30-minute intervals (0 hours [08:30], 0.5 hours, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours and 4 hours). Subjective appetite ratings will be measured at 30-minute intervals (0 hours [08:30], 0.5 hours, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours and 4.5 hours). Participants will complete the Burghart ODOFIN Sniffin' Sticks smell test and the Burghart ODOFIN taste strips test at three time points during the trials (0 hours [08:30], 1.5 hours and 4 hours). Participants will rest for the duration of the trials except for performing 1 hour of treadmill exercise (walking/jogging) at 60% of their peak oxygen uptake (calculated from the pre-visit) between 0.5 to 1.5 hours (09:00-10:00) in the exercise trial. Expired air samples will be collected during exercise and for 30 minutes during the rest trial to calculate net energy expenditure and substrate oxidation. At 2.5 hours (11:00), an ad libitum lunch consisting of a homogeneous meal containing pasta, tomato sauce, and olive oil (72% carbohydrate, 12% protein, 16% fat, 6.5 kJ per gram of food) will be provided for 30 minutes (until 3 hours).

The MRI visit will take place after an overnight fast of at least 10 hours and will involve a 45 minute scanning protocol. Structural MRI and functional MRI (fMRI) scans will be performed on a GE 3.0 T Discovery MR750w scanner using a 32 channel head coil. Two fMRI scans will be performed (1) during the presentation of food and non-food cues and (2) for an equivalent duration whilst participants are not looking at food and non-food cues.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 - 24.9 kg/m2 and a waist circumference of ≤ 88 cm for women, and ≤ 102 cm for men or a BMI between 25 - 40 kg/m2 and a waist circumference of > 88 cm for women, and > 102 cm for men. BMI and waist circumference thresholds vary amongst ethnicities. People with a South Asian, Chinese, other Asian, Middle Eastern, Black African or African-Caribbean family background are prone to central adiposity and their cardiometabolic risk occurs at a lower BMI. Therefore, the following BMI and waist circumference thresholds will be applied for people of South Asian, other Asian, Black African and African-Caribbean ethnicity: (1) BMI 18.5 kg/m2 to 23 kg/m2 and waist circumference of < 90 cm for men and < 80 cm for women; (2) BMI 23.1 kg/m2 to 40 kg/m2 and waist circumference of ≥ 90 cm for men and ≥ 80 cm for women.
* Normally consumes three meals a day
* Able to walk continuously for 1 hour on a treadmill
* Weight stable for 3 months (< 3kg change in weight)
* Regular menstrual cycle for the last 6 months (people taking the combined contraceptive pill are eligible for the study)
* Able to undergo a 45-minute MRI scan

Exclusion Criteria:

* Smokers (vaping is considered smoking in this study)
* Known medical conditions (e.g. diabetes, heart condition)
* Taking any medication which may affect the study outcomes (e.g. liraglutide, semaglutide, insulin, steroids, anti-psychotics)
* Clinically diagnosed eating disorder
* Previous bariatric surgery (e.g. gastric bypass, gastric band, sleeve gastrectomy)
* Food allergies or intolerances, or severe dislikes to study foods
* Pregnant or breastfeeding
* Have recently donated blood (within eight weeks of visits 2 and 3).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-05 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Concentration of Oxyntomodulin | Blood samples to measure oxyntomodulin are collected at 30-minute intervals (0 hours [08:30], 0.5 hours, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours and 4 hours) in each trial.
  Plasma blood samples

SECONDARY OUTCOMES:
Concentration of Acylated Ghrelin | Blood samples to measure acylated ghrelin are collected at 30-minute intervals (0 hours [08:30], 0.5 hours, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours and 4 hours) in each trial.
  Acylated Ghrelin. Blood plasma sample.
Concentration of Leptin | Blood samples to measure leptin are collected at 0 hours [08:30] in each trial.
  Blood plasma sample.
Concentration of Glucagon-like peptide 1 | Blood samples to measure GLP-1 are collected at 30-minute intervals (0 hours [08:30], 0.5 hours, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours and 4 hours) in each trial.
  Glucagon-like peptide 1 (GLP-1). Blood plasma sample.
Concentration of Peptide YY | Blood samples to measure PYY are collected at 30-minute intervals (0 hours [08:30], 0.5 hours, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours and 4 hours) in each trial.
  Peptide YY (PYY) plasma blood sample
Concentration of Glucose | Blood samples to measure glucose are collected at 30-minute intervals (0 hours [08:30], 0.5 hours, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours and 4 hours) in each trial.
  Blood plasma sample
Visual analogue score (VAS) for subjective appetite | VAS is measured at 30-minute intervals (0 hours [08:30], 0.5 hours, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours and 4.5 hours) in each trial.
  Participants subjective appetite sensations are assessed using 100mm visual analogue scales to measure four appetite constructs: 'hunger', 'fullness', 'satiety' and 'prospective food consumption'.
Energy intake | The ad libitum pasta meal is provided at 2.5 hours (11:00)
  (kcal). A large bowl containing an amount of pasta in excess of expected consumption is presented to participants for 30 minutes. They are instructed to self-serve and to stop eating when they reach volitional satiation. The remaining food is weighed and subtracted from the known quantity initially presented to calculate ad libitum energy intake.
Gustatory perceptions | The taste tests will take place at three time points during the trials: 0 hours [08:30], 1.5 hours and 4 hours.
  The Burghart ODOFIN taste strips test is used to evaluate participant's ability to detect different taste sensations. It assesses the sensitivity of a person's taste buds to various taste qualities, including sweet, salty, sour, bitter, and umami (savoury) and some taste strips may have no taste at all (neutral). The paper strips are placed in the middle of the anterior tongue and the participant will be asked to identify the taste. Participants are asked to take a sip of water between each paper strip.
Olfactory perceptions | The smell tests will take place at three time points during the trials: 0 hours [08:30], 1.5 hours and 4 hours.
  The Burghart ODOFIN Sniffin' Sticks smell test is used to evaluate the person's ability to detect, identify, and differentiate various odours. The test involves presenting a series of different odours in the form of sniff pens. The participant will be asked to sniff each pen and then identify each odour from a card which is presented to them.
Task-based fMRI | 45-minute scan at baseline
  Brain responses to visual food cues assessed during the presentation of food and non-food images
Resting state fMRI | 45-minute scan at baseline
  Functional activity of the brain assessed at rest.

CONTACTS AND LOCATIONS:
Overall Officials: David J Stensel, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available to researchers upon request.